CLINICAL TRIAL: NCT07179406
Title: The Effect of Spinal Cord Stimulators on Restless Leg Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Marshall Holland, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300014915; UAB (Other: UAB)
Record Dates: First submitted 2025-08-28; First posted 2025-09-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Restless Leg Syndrome (RLS); Spinal Cord Stimulation (SCS)
Keywords: SCS; Spinal Cord Stimulation; RLS; Restless Leg Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — H-Reflex; Evoked Potentials, Somatosensory; Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Assessments and questionnaires only (Active Comparator): Complete questionnaires on RLS and pain
  Stimulation:
  H-reflex - A small electrical stimulus is provided to the leg and foot area and a measurement of the stimulus is taken by the EEG electrodes.
  Somatosensory evoked potential (SSEP) - A small electrical stimulus is provided to a nerve on the body and measured at several places along the nervous system (spinal cord, brain, etc.) with the EMG and EEG electrodes.
  Vibratory Electrophysiological Response Potential (ERP) - stimulation of the ankle with vibration sensations using a device like a buzzer and recording of body's responses using the EEG and/or EMG electrodes.
  Transcranial Magnetic Stimulation (TMS) - A small magnetic pulse is used to provide a small amount of electrical stimulation to nervous system. The EEG and/or EMG electrodes will be used to measure body's reaction.
  Interventions: Other: H-Reflex; Other: Somatosensory evoked potential (SSEP); Other: Vibratory Electrophysiological Response Potential (ERP); Other: Transcranial Magnetic Stimulation (TMS)
- Arm 2: Off-on-off (Active Comparator): Participants will turn OFF their SCS at least 48 hours prior to the visit. The assessments listed in Arm 1 will be performed and the SCS will be turned ON for at least 60 minutes before repeating the assessments. Participants may repeat the questionnaires during this waiting period.
  Finally, the SCS is turned OFF again, this time for at least 30 minutes before repeating the assessments, except for the h-reflex, which will not be needed again. As with before, participants can complete the questionnaires during this waiting period.
  Interventions: Other: H-Reflex; Other: Somatosensory evoked potential (SSEP); Other: Vibratory Electrophysiological Response Potential (ERP); Other: Transcranial Magnetic Stimulation (TMS); Other: Spinal Cord Stimulator (SCS) manipulation
- Arm 3: Off-on-off post-op (Active Comparator): Participants will perform the same procedures as those in Arm 2, but only after 2-3 weeks from receiving a permanent SCS.
  Interventions: Other: H-Reflex; Other: Somatosensory evoked potential (SSEP); Other: Vibratory Electrophysiological Response Potential (ERP); Other: Transcranial Magnetic Stimulation (TMS); Other: Spinal Cord Stimulator (SCS) manipulation
- Arm 4: On-off-on (Active Comparator): Participants will have their SCS on for at least 48 hours prior to the visit. The assessments listed in Arm 1 will be performed and the SCS will be turned Off for at least 60 minutes before repeating the assessments. Participants may repeat the questionnaires during this waiting period.
  Finally, the SCS is turned On again, this time for at least 30 minutes before repeating the assessments, except for the h-reflex, which will not be needed again. As with before, participants can complete the questionnaires during this waiting period.
  Interventions: Other: H-Reflex; Other: Somatosensory evoked potential (SSEP); Other: Vibratory Electrophysiological Response Potential (ERP); Other: Transcranial Magnetic Stimulation (TMS); Other: Spinal Cord Stimulator (SCS) manipulation

INTERVENTIONS:
Other: H-Reflex — H-reflex - A small electrical stimulus is provided to the leg and foot area and a measurement of the stimulus is taken by the EEG electrodes.
Other: Somatosensory evoked potential (SSEP) — A small electrical stimulus is provided to a nerve on the body and measured at several places along the nervous system (spinal cord, brain, etc.) with the EMG and EEG electrodes.
Other: Vibratory Electrophysiological Response Potential (ERP) — stimulation is provided to the ankle with vibration sensations using a device like a buzzer and the recording of the body's responses using the EEG and/or EMG electrodes.
Other: Transcranial Magnetic Stimulation (TMS) — A small magnetic pulse is used to provide a small amount of electrical stimulation to the nervous system. The EEG and/or EMG electrodes will be used to measure the body's reaction.
Other: Spinal Cord Stimulator (SCS) manipulation — Spinal cord stimulator will be turned on/off
  Arms: Arm 2: Off-on-off; Arm 3: Off-on-off post-op; Arm 4: On-off-on

SUMMARY:
This study aims to evaluate neurophysiological responses and symptom changes in individuals with Restless Legs Syndrome (RLS) and/or chronic pain. Participants will undergo standard clinical assessments including EEG, EMG, h-reflex, SSEP, ERP, and TMS under varying SCS conditions.The study involves 4 arms. Arm 1 are individuals diagnosed with RLS and Healthy Controls. Arm 2 are individuals diagnosed with RLS and have an existing SCS. Arm 3 are individuals diagnosed with RLS and scheduled to receive a SCS. Arm 4 are individuals with chronic pain and have a SCS, but no diagnosis of RLS.

ELIGIBILITY:
Inclusion Criteria:

* Has Restless Leg Syndrome
* No major changes in RLS medications in past 4 weeks
* Willing and able to comply with study protocol
* Healthy Controls - No RLS diagnosis
* Ability to provide informed consent

Exclusion Criteria:

* Any mental or physical limitation that would prevent completing any of the studies
* Currently using another device to treat RLS
* Unable or unwilling to comply with study protocols
* Other medical condition that would put the subject at risk as determined by the investigator
* Pregnant, breastfeeding, or trying to become pregnant
* Currently participating or planning to participate in any other investigational clinical evaluation during the study period that may, in the opinion of the investigator, affect RLS
* One or more of the following diseases: spinal cord injury, severe peripheral neuropathy or radiculopathy, severe psychiatric or cognitive disorder that may interfere with participation of the study, history of drug or alcohol abuse within the past year, epilepsy or seizure disorder, current active or chronic infection other than the common cold, malignancy within the past 5 years (not including basal cell or squamous cell skin cancer), severe movement disorder (i.e. Parkinson's disease), deep vein thrombosis, or multiple sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in H-reflex neurophysiological activity in response to Spinal Cord Stimulation (SCS) | Up to 3 Weeks after consent to the study
Changes in Somatosensory Evoked Potential (SSEP) activity in response to Spinal Cord Stimulation (SCS) | Up to 3 Weeks after consent to the study
Changes in Vibratory Electrophysiological Response Potential (ERP) activity in response to Spinal Cord Stimulation (SCS) | Up to 3 Weeks after consent to the study
Changes in Transcranial Magnetic Stimulation (TMS) activity in response to Spinal Cord Stimulation (SCS) | Up to 3 Weeks after consent to the study

SECONDARY OUTCOMES:
Changes in self-reported RLS symptoms via International Restless Legs Syndrome (IRLSS) Questionnaire | Up to 3 Weeks after consent to the study
Changes in self-reported RLS symptoms via RLS-6 Questionnaire | Up to 3 Weeks after consent to the study
Changes in self-reported pain symptoms via Promis Questionnaire | Up to 3 Weeks after consent to the study
Changes in self-reported pain symptoms via PainDetect Questionnaire | Up to 3 Weeks after consent to the study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States